CLINICAL TRIAL: NCT03453619
Title: A Phase 2 Study to Evaluate the Safety and Biologic Activity of APL- 2 in Patients With IgA Nephropathy, Lupus Nephritis, Primary Membranous Nephropathy, or C3 Glomerulopathy (C3 Glomerulonephritis and Dense Deposit Disease)
Brief Title: Phase II Study Assessing Safety and Efficacy of APL-2 in Glomerulopathies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-201
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-07

CONDITIONS: IgA Nephropathy; Lupus Nephritis; Membranous Nephropathy; C3 Glomerulonephritis; Dense Deposit Disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Lupus Nephritis; Glomerulonephritis, Membranous; Glomerulonephritis, Membranoproliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APL-2 (Experimental): Open Label, Study Drug, APL-2
  Interventions: Drug: APL-2

INTERVENTIONS:
Drug: APL-2 — APL-2 administered as a daily subcutaneous infusion for 48 weeks

SUMMARY:
This is a Phase II trial assessing the safety and preliminary efficacy of daily APL-2 subcutaneous infusion administered for 16 weeks with a 6 month safety follow up, in patients with glomerulopathies

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years of age at screening (16 years of age for C3G), able to provide written informed consent, and able to understand and comply with all scheduled procedures and other requirements of the study by the opinion of Principal Investigator (PI)
* Patients must have a diagnosis of IgAN, LN, Primary MN, or C3G confirmed by renal biopsy and required measurements performed prior to study participation

  * IgAN: Prior biopsy results for C3 and C4d staining should be made available
  * LN: Diagnostic biopsy showing proliferative focal, diffuse, or membranous lesions (Class III, IV or V, respectively) by renal biopsy. Subject should have either a biopsy in the last 6 months, or evidence of disease activity (nephritic changes on urinalysis or nephrotic changes)
  * Primary MN: PLA2R positive titer plus nephrotic range proteinuria (defined as uPCR >2350 mg/g)
  * C3G plus one of the following: Low serum C3 level or historical renal biopsy within the last 3 years
* Have proteinuria >750 mg/g (calculated by uPCR on 24 hour urine collection) collected during the first screening visit (Visit 3a).
* eGFR≥30mL/min/1.73 m2 calculated by CKD-EPI creatinine equation at screening visit 3a and currently not on dialysis
* Must have stable or worsening renal disease, on stable and optimized treatment, in the opinion of the PI, for at least 2 months prior to the first dose of APL-2 (Visit 4); treatments may include, but are not limited to, immunosuppressive agents, anti-hypertensives and/or anti-proteinurics.
* Willing to receive vaccinations against Neisseria meningitidis at least 2 weeks prior to dosing on Day 1 with a booster on Day 56 (for both vaccinations) and Pneumococcal and Hib vaccines at least 2 weeks prior to dosing on Day 1.

Exclusion Criteria:

* Absolute neutrophil count <1000 cells/mm3 at screening Visits 3a and 3b
* ALT or AST >3.0 x the upper limit of normal at screening Visits 3a and 3b
* Previous treatment with APL-2
* History of solid organ transplant
* Diagnosis of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection, or positive serology at screening Visits 3a and 3b (previous HBV or HCV diagnosis cleared by treatment is allowed)
* Renal disease secondary to another condition (e.g. infection, malignancy, monoclonal gammopathy, or a medication)
* Presence or suspicion of active bacterial or viral infection or severe recurrent bacterial infections
* Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedure within 30 days prior to screening period
* Unwillingness to receive or intolerant of SC infusions of study medication or known allergy to ingredients in APL-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2023-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - HealthONE Physician Care, Rocky Mountain Hospital for Children, Denver, Colorado
  - Washington Nephrology Associates, Washington D.C., District of Columbia
  - Horizon Research Group, Coral Gables, Florida
  - Emory University, Atlanta, Georgia
  - American Research LLC, Jeffersonville, Indiana
  - Northwest Louisiana Nephrology LLC, Shreveport, Louisiana
  - Washington Nephrology Associates, Takoma Park, Maryland
  - Clinical Research Consultants, Kansas City, Missouri
  - Davita Clinical Research, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Southeastern Nephrology Associates, Wilmington, North Carolina
  - University Clinical Health, Memphis, Tennessee
  - Washington Nephrology Associates, Alexandria, Virginia
  - Davita Clinical Research, Chesapeake, Virginia
  - Milwaukee Nephrologists, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Budge KL, Verlato A, Bin S, Salem FE, Perin L, La Manna G, Zaza G, Fiaccadori E, Cantarelli C, Cravedi P. Decay-Accelerating Factor Restrains Complement Activation and Delays Progression of Murine cBSA-Induced Membranous Nephropathy. Kidney360. 2023 Jun 1;4(6):e769-e776. doi: 10.34067/KID.0000000000000122. Epub 2023 Apr 8. PMID 37036696

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective Phase 2, open-label study was conducted in subjects clinically diagnosed with immunoglobulin A nephropathy (IgAN), lupus nephritis (LN), primary membranous nephropathy (PMN), or C3 glomerulopathy (C3G) between 26 February 2018 and 25 August 2023.
Pre-assignment Details: The study consisted of 2 parts: Part A (core study phase; 48 weeks) and Part B (long-term extension phase; until pegcetacoplan was commercially available for the disease under treatment). Subjects were screened within 4 weeks prior to the start of dosing on Day 1. A total of 21 subjects were enrolled in this study.
Groups:
- IgAN Subjects: Subjects diagnosed with IgAN received pegcetacoplan 360 milligram (mg) subcutaneous (SC) infusion once daily up to 48 weeks in Part A and eligible subjects entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
- LN Subjects: Subjects diagnosed with LN received pegcetacoplan 360 mg SC infusion once daily up to 48 weeks in Part A and eligible subjects entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
- PMN Subjects: Subjects diagnosed with PMN received pegcetacoplan 360 mg SC infusion once daily up to 48 weeks in Part A and eligible subjects entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
- C3G Subjects: Subjects diagnosed with C3G received pegcetacoplan 360 mg SC infusion once daily up to 48 weeks in Part A and eligible subjects entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
Period: Core Study (Part A)
Arm/Group | IgAN Subjects | LN Subjects | PMN Subjects | C3G Subjects
Started | 6 | 2 | 5 | 8
Completed (Completed Part A.) | 4 | 1 | 1 | 7
Not Completed | 2 | 1 | 4 | 1
Not completed — Physician Decision | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 1
Not completed — Other | 0 | 1 | 0 | 0
Period: Long-Term Extension (Part B)
Arm/Group | IgAN Subjects | LN Subjects | PMN Subjects | C3G Subjects
Started (Subjects rolled over to Part B.) | 4 | 1 | 0 (Subject completed Part A but didn't enter the Part B of study.) | 7
Completed (Completed Part B.) | 2 | 0 | 0 | 5
Not Completed | 2 | 1 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population included all subjects who received at least 1 dose of pegcetacoplan.
Groups:
- IgAN Subjects: Subjects diagnosed with IgAN received pegcetacoplan 360 mg SC infusion once daily up to 48 weeks in Part A and eligible subjects entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
- Total: Total of all reporting groups
Arm/Group | IgAN Subjects | LN Subjects | PMN Subjects | C3G Subjects | Total
Number analyzed (Participants) | 6 | 2 | 5 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (14.18) | 44.5 (10.61) | 62.2 (7.43) | 22.5 (8.65) | 40.5 (18.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 5 | 7
  Male | 5 | 2 | 4 | 3 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 4 | 0 | 4 | 6 | 14
  Other | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline in Proteinuria at Week 48
Description: Change from baseline in proteinuria was assessed based on urinary protein-to-creatinine ratio (uPCR). Baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug.
Time Frame: Baseline (Day 1) and Week 48
Population: The intent-to-treat (ITT) population included all subjects who received at least 1 dose of pegcetacoplan. Only subjects analyzed at baseline and Week 48 are reported.
Measure: Mean (95% Confidence Interval); unit: ratio
Groups:
- Part A: IgAN Subjects: Subjects diagnosed with IgAN received pegcetacoplan 360 mg SC infusion once daily up to 48 weeks in Part A.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
- Part A: LN Subjects: Subjects diagnosed with LN received pegcetacoplan 360 mg SC infusion once daily up to 48 weeks in Part A.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
- Part A: PMN Subjects: Subjects diagnosed with PMN received pegcetacoplan 360 mg SC infusion once daily up to 48 weeks in Part A.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
- Part A: C3G Subjects: Subjects diagnosed with C3G received pegcetacoplan 360 mg SC infusion once daily up to 48 weeks in Part A.
  Subjects were able to switch over to twice-weekly dosing with pegcetacoplan 1080 mg, as early as Week 24, but no later than the entrance into Part B.
Arm/Group | Part A: IgAN Subjects | Part A: LN Subjects | Part A: PMN Subjects | Part A: C3G Subjects
Number analyzed (Participants) | 5 | 1 | 1 | 7
ratio | -0.1364 [-1.0641 to 0.7913] | 0.3560 [NA to NA] — The 95% confidence interval (CI) couldn't be determined as only 1 subject was analyzed. | 0.3430 [NA to NA] — The 95% CI couldn't be determined as only 1 subject was analyzed. | -2.0347 [-3.9033 to -0.1662]

2. Secondary Outcome: Parts A and B: Change From Baseline in Serum Complement 3 (C3) Levels at Week 48 of Part A and Week 168 of Part B
Description: Blood samples were collected to measure serum C3 levels. Part A baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug. Part B baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug during Part B.
Time Frame: Part A: Baseline (Day 1) and Week 48; Part B: Baseline (Part A, Week 48) and Week 168
Population: The ITT population included all subjects who received at least 1 dose of pegcetacoplan. Only subjects analyzed at baseline and specific timepoints are reported.
Measure: Mean (95% Confidence Interval); unit: milligram per deciliter
Groups:
- Part B: IgAN Subjects: Eligible subjects diagnosed with IgAN entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
- Part B: LN Subjects: Eligible subjects diagnosed with LN entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
- Part B: C3G Subjects: Eligible subjects diagnosed with C3G entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
Arm/Group | Part A: IgAN Subjects | Part A: LN Subjects | Part A: PMN Subjects | Part A: C3G Subjects | Part B: IgAN Subjects | Part B: LN Subjects | Part B: C3G Subjects
Number analyzed (Participants) | 6 | 0 | 1 | 7 | 2 | 0 | 4
milligram per deciliter | 153.17 [27.94 to 278.39] |  | 324.00 [NA to NA] — The 95% confidence interval (CI) couldn't be determined when only 1 participant was analyzed. | 194.43 [109.45 to 279.41] | -74.00 [-506.01 to 358.01] |  | -48.50 [-214.73 to 117.73]

3. Secondary Outcome: Parts A and B: Change From Baseline in Alternative Pathway Hemolytic Assay (AH50) Activity at Week 48 of Part A and Week 168 of Part B
Description: Blood samples were collected to measure AH50 activity. Part A baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug. Part B baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug during Part B.
Time Frame: Part A: Baseline (Day 1) and Week 48; Part B: Baseline (Part A, Week 48) and Week 168
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units per milliliter
Arm/Group | Part A: IgAN Subjects | Part A: LN Subjects | Part A: PMN Subjects | Part A: C3G Subjects | Part B: IgAN Subjects | Part B: LN Subjects | Part B: C3G Subjects
Number analyzed (Participants) | 6 | 0 | 1 | 6 | 2 | 0 | 4
units per milliliter | -17.3 [-71.0 to 36.3] |  | -48.0 [NA to NA] — The 95% CI couldn't be determined when only 1 participant was analyzed. | 4.0 [-59.7 to 67.7] | 9.0 [-16.4 to 34.4] |  | 27.0 [-89.7 to 143.7]

4. Secondary Outcome: Parts A and B: Change From Baseline in C3a Concentrations at Week 48 of Part A and Week 168 of Part B
Description: Blood samples were collected to measure C3a concentrations. Part A baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug. Part B baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug during Part B.
Time Frame: Part A: Baseline (Day 1) and Week 48; Part B: Baseline (Part A, Week 48) and Week 168
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: microgram per liter
Arm/Group | Part A: IgAN Subjects | Part A: LN Subjects | Part A: PMN Subjects | Part A: C3G Subjects | Part B: IgAN Subjects | Part B: LN Subjects | Part B: C3G Subjects
Number analyzed (Participants) | 6 | 0 | 1 | 5 | 2 | 0 | 4
microgram per liter | 1283.93 [-1963.09 to 4530.95] |  | 56.30 [NA to NA] — The 95% CI couldn't be determined when only 1 participant was analyzed. | 55.16 [-173.33 to 283.65] | -10.00 [-41.77 to 21.77] |  | -100.65 [-361.20 to 159.90]

5. Secondary Outcome: Parts A and B: Change From Baseline in Serum Albumin Levels at Week 48 of Part A and Week 168 of Part B
Description: Blood samples were collected to measure serum albumin levels. Part A baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug. Part B baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug during Part B.
Time Frame: Part A: Baseline (Day 1) and Week 48; Part B: Baseline (Part A, Week 48) and Week 168
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: gram per deciliter
Arm/Group | Part A: IgAN Subjects | Part A: LN Subjects | Part A: PMN Subjects | Part A: C3G Subjects | Part B: IgAN Subjects | Part B: LN Subjects | Part B: C3G Subjects
Number analyzed (Participants) | 6 | 0 | 2 | 7 | 2 | 0 | 3
gram per deciliter | -0.17 [-0.81 to 0.48] |  | 0.20 [-6.15 to 6.55] | 0.59 [-0.29 to 1.46] | -0.30 [-6.65 to 6.05] |  | -0.53 [-3.60 to 2.53]

6. Secondary Outcome: Parts A and B: Number of Subjects With Complete Clinical Remission at Week 48 of Part A and Week 168 of Part B
Description: The complete clinical remission was defined as normalization of proteinuria as defined by <200 mg/g uPCR.
Time Frame: Part A: Week 48; Part B: Week 168
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: IgAN Subjects | Part A: LN Subjects | Part A: PMN Subjects | Part A: C3G Subjects | Part B: IgAN Subjects | Part B: LN Subjects | Part B: C3G Subjects
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 2 | 0 | 4
Participants
  <200 | 0 | 0 | 0 | 0 | 0 |  | 1
  >=200 | 5 | 1 | 1 | 7 | 2 |  | 3

7. Secondary Outcome: Parts A and B: Number of Subjects With Stabilization or Improvement in Estimated Glomerular Filtration Rate (eGFR) From Baseline at Week 48 of Part A and Week 168 of Part B
Description: The eGFR stabilization or improvement was defined as an eGFR value that was no more than a 25% decrease relative to baseline. Part A baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug. Part B baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug during Part B.
Time Frame: Part A: Baseline (Day 1) and Week 48; Part B: Baseline (Part A, Week 48) and Week 168
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: IgAN Subjects | Part A: LN Subjects | Part A: PMN Subjects | Part A: C3G Subjects | Part B: IgAN Subjects | Part B: LN Subjects | Part B: C3G Subjects
Number analyzed (Participants) | 6 | 0 | 2 | 7 | 2 | 0 | 3
Participants
  Stable GFR: no more than 25% (+/-) change | 3 | 0 | 1 | 5 | 2 |  | 3
  Improvement in GFR: >25% increase | 0 | 0 | 0 | 1 | 0 |  | 0
  Worsening of GFR: >25% decrease | 3 | 0 | 1 | 1 | 0 |  | 0

8. Primary Outcome: Part B: Change From Baseline in Proteinuria at Week 168
Description: Change from baseline in proteinuria was assessed based on uPCR. Baseline was defined as the most recent non-missing measurement prior to or on the first administration of study drug during Part B.
Time Frame: Baseline (Part A, Week 48) and Week 168
Population: The ITT population included all subjects who received at least 1 dose of pegcetacoplan. Only subjects analyzed at baseline and Week 168 are reported.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: IgAN Subjects | Part B: LN Subjects | Part B: C3G Subjects
Number analyzed (Participants) | 2 | 0 | 4
ratio | -0.3385 [-3.8264 to 3.1494] |  | 0.9718 [-4.7933 to 6.7368]

ADVERSE EVENTS:
Time Frame: TEAE data is reported from first dose of study drug (Day 1) up to 56 days after the last dose of study drug, up to approximately 1745 days.
Description: The Safety population included all subjects who received at least 1 dose of pegcetacoplan. MedDRA version for Part A was 23.0 and Part B was 26.0.
Groups:
- Part B: PMN Subjects: Eligible subjects diagnosed with PMN entered Part B to continue to receive pegcetacoplan 360 mg SC infusion until it was commercially available for the disease under treatment.
Arm/Group | Part A: IgAN Subjects | Part A: LN Subjects | Part A: PMN Subjects | Part A: C3G Subjects | Part B: IgAN Subjects | Part B: LN Subjects | Part B: PMN Subjects | Part B: C3G Subjects
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/5 | 0/8 | 0/4 | 0/1 | 0/0 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 4/5 | 0/8 | 1/4 | 1/1 | 0/0 | 1/7
Other Adverse Events (participants affected / at risk) | 5/6 | 1/2 | 5/5 | 8/8 | 4/4 | 1/1 | 0/0 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: IgAN Subjects (N=6) | Part A: LN Subjects (N=2) | Part A: PMN Subjects (N=5) | Part A: C3G Subjects (N=8) | Part B: IgAN Subjects (N=4) | Part B: LN Subjects (N=1) | Part B: PMN Subjects (N=0) | Part B: C3G Subjects (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 1
End-stage renal disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: IgAN Subjects (N=6) | Part A: LN Subjects (N=2) | Part A: PMN Subjects (N=5) | Part A: C3G Subjects (N=8) | Part B: IgAN Subjects (N=4) | Part B: LN Subjects (N=1) | Part B: PMN Subjects (N=0) | Part B: C3G Subjects (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | NA | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | NA | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | NA | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 1 | 1 | NA | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | NA | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | NA | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | NA | 1
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0
Injection site discomfort (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | NA | 0
Injection site erythema (General disorders) | 2 | 0 | 1 | 1 | 0 | 0 | NA | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 1
Injection site pruritus (General disorders) | 0 | 0 | 1 | 2 | 1 | 0 | NA | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | NA | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Injury associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 2
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | NA | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | NA | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | NA | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | NA | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 2 | 0 | 0 | NA | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | NA | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Acoustic shock (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | NA | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Skin procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 2
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Cystatin C increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 1
Hyperphagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Chronic kidney disease-mineral and bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | NA | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 3 | 0 | 1 | NA | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | NA | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | 0
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | NA | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Vaginal odour (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | NA | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | 0
Acne cystic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 1
Fracture treatment (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Polypectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03453619/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03453619/SAP_001.pdf